CLINICAL TRIAL: NCT03581370
Title: Comparison of Short Infusion Versus Prolonged Infusion of Ceftolozane-tazobactam Among Patients with Ventilator Associated-pneumonia to Pseudomonas Aeruginosa in Intensive Care Units
Brief Title: Short Infusion Versus Prolonged Infusion of Ceftolozane-tazobactam Among Patients with Ventilator Associated-pneumonia
Acronym: CEFTOREA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 31/17/0334; 2018-000059-42 (EudraCT Number)
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Pneumonia; Pseudomonas aeruginosa; pharmacokinetics
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia; Pseudomonas Infections | interventions — ceftolozane, tazobactam drug combination; Powders

STUDY DESIGN:
Intervention Model Description: The patient will be randomized either in the 4-hours or in the 1-hour infusion group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 hour infusion (Active Comparator): The first group corresponds to 1-hour infusion : First administration of ceftolozane-tazobactam with 2000 mg by infusion for 60 minutes every 8 hours.
  24h after this first administration, 7 blood samples will be collected at Hour 24, Hour 25, Hour 26, Hour 28, Hour 30, Hour 32 and Hour 48.
  Interventions: Drug: 1 hour infusion
- 4 hours infusion (Experimental): The second group corresponds to 4-hours infusion: First administration of ceftolozane-tazobactam with 2000 mg by infusion for 4 hours every 8 hours. 24h after this first administration, 7 blood samples will be collected at Hour 24, Hour 25, Hour 26, Hour 28, Hour 30, Hour 32 and Hour 48.
  .
  Interventions: Drug: 4 hours infusion

INTERVENTIONS:
Drug: 1 hour infusion — Intravenous administration of ceftolozane-tazobactam (ZERBAXA®) : 2000 mg by infusion for 60 minutes every 8 hours.
  Other Names: Zerbaxa 1 g/0.5 g powder
  Arms: 1 hour infusion
Drug: 4 hours infusion — Intravenous administration of ceftolozane-tazobactam (ZERBAXA®) : 2000 mg by infusion for 4 hours every 8 hours
  Other Names: Zerbaxa 1 g/0.5 g powder
  Arms: 4 hours infusion

SUMMARY:
The main objective of this study is to compare the median exposures at pharmacokinetic equilibrium of the two modalities of administration: 4-hours infusion of ceftolozane-tazobactam at a dosage of 2 gram three times a day vs 1-hour infusion of 2 gram three times a day.

DETAILED DESCRIPTION:
Intensive care unit patients with ventilator associated-pneumonia often develop severe and rapidly life threatening Gram-negative Bacillus infections. Moreover, they present pathophysiological disturbances responsible for major pharmacokinetic changes (volume of distribution and glomerular filtration) which may lead to drugs under-exposure. Any delay in management or inadequate antibiotic therapy can have serious consequences in terms of prognosis. The association ceftolozane-tazobactam is an alternative to carbapenems in documented infections. Ceftolozane is a new cephalosporin, marketed, in combination with tazobactam (beta-lactamase inhibitor) under the name ZERBAXA®. ZERBAXA® is active on Gram-negative Bacillus, including Pseudomonas aeruginosa.

This is a prospective, randomized, open pharmacokinetic/pharmacodynamic study that compares two modalities of administration of a novel antibiotic, ZERBAXA® ceftolozane-tazobactam, by 4-hours infusion at the dosage of 2 gram three times a day vs. 1-hour infusion at the dosage of 2 g three times a day, among patients with ventilator associated-pneumonia to Pseudomonas aeruginosa.

The patient will be randomized either in the 4-hours or in the 1-hour infusion group. Follow up visits are daily for any intensive care patient. Those provided for biomedical research are carried out during the treatment period, at Day 15 and Day 28. For the pharmacokinetic study, 7 blood samples will be collected from 24 hours to 48 hours after the first ZERBAXA® administration.

ELIGIBILITY:
inclusion criteria

* patients with ventilator associated-pneumonia to Pseudomonas aeruginosa
* patients hospitalized in intensive care units
* Pseudomonas aeruginosa susceptible to ceftolozane-tazobactam
* Simplified Acute Physiological Score II (SAPS II () > 20
* Expected duration of survival > 7 days
* Informed consent of the patient or, failing that, the patient's close or trustworthy person
* Affiliated to a social security scheme or equivalent

Non inclusion criteria:

* history of allergy to one of the two molecules
* history of allergy to betalactamines
* Strain Isolated resistant to Ceftolozane-Tazobactam combination
* Renal insufficiency with a glomerular filtration rate evaluated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) < 50 ml/min
* Patient on dialysis or under continuous hemodiafiltration
* pregnant or nursing women
* patient benefiting from a system of legal protection for adults
* patient with active immunodepression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Time that the concentration spends above 5 Minimum inhibitory Concentration (T>5*MIC) | Time between two administrations (8 hours)
  The primary endpoint is the time that the concentration spends above 5* Minimum inhibitory Concentration, expressed as a percentage of the time interval between two administrations. The T>5* Minimum inhibitory Concentration will be determined for each patient from the concentration profile measured over an 8-hour post-administration interval. Since protein binding is low (<20%), the total concentration (sum of free form and plasma protein bound) will be used as a marker for free concentration. Therefore, the T>5* Minimum inhibitory Concentration will be calculated from the total concentrations. Our study will focus on only Pseudomonas aeruginosa Pneumonia acquired under mechanical ventilation with a critical Minimum inhibitory Concentration of 4 mg/l, T>5* Minimum inhibitory Concentration will then correspond to a residual serum concentration of 20 mg/l.

SECONDARY OUTCOMES:
Percentage of patients with concentrations greater than 5*Minimum inhibitory Concentration | Time between two administrations (8 hours)
  The percentage of patients with concentrations greater than 5*Minimum inhibitory Concentration over an 8-hour post administration interval.
Bactericidal rate | at Day 10
  Bactericidal rate obtained in vitro using the Hollow Fiber device. This rate is determined for broncho-alveolar concentrations estimated in patients with pneumonia acquired during ventilation
Percentage of patients recovering at the end of the treatment period | at Day 10
  Number of patients recovering in relation to the total number of patients
Percentage of patients failing at the end of the treatment period | at Day 10
  Number of patients failing in relation to the total number of patients
Number of days without artificial ventilation | at Day 28
  The number of days without artificial ventilation
The duration of hospitalization | at Day 28
  the duration of hospitalization in number of day
Survival at D28 | at Day 28
  survival in number of patient alive
The alveolar concentration of Ceftolozane-Tazobactam | between 24 hour and 48 hour after time 0
  The alveolar concentration of Ceftolozane-Tazobactam from a sample of the alveolar fluid produced by bronchial fibroscopy between the 24th hour and the 48th hour
Evaluation of the serious adverse events | Day 28
  Evaluation of the serious adverse events at the doses and regimen recommended in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie RUIZ, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service Réanimation Polyvalente - CHU Rangueil, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colomb-Cotinat M, Lacoste J, Brun-Buisson C, Jarlier V, Coignard B, Vaux S. Estimating the morbidity and mortality associated with infections due to multidrug-resistant bacteria (MDRB), France, 2012. Antimicrob Resist Infect Control. 2016 Dec 12;5:56. doi: 10.1186/s13756-016-0154-z. eCollection 2016. PMID 27999665
- [Background] Vincent JL, Bassetti M, Francois B, Karam G, Chastre J, Torres A, Roberts JA, Taccone FS, Rello J, Calandra T, De Backer D, Welte T, Antonelli M. Advances in antibiotic therapy in the critically ill. Crit Care. 2016 May 17;20(1):133. doi: 10.1186/s13054-016-1285-6. PMID 27184564
- [Background] Gelfand MS, Cleveland KO. Ceftolozane/Tazobactam Therapy of Respiratory Infections due to Multidrug-Resistant Pseudomonas aeruginosa. Clin Infect Dis. 2015 Sep 1;61(5):853-5. doi: 10.1093/cid/civ411. Epub 2015 May 28. No abstract available. PMID 26021991
- [Background] Monogue ML, Pettit RS, Muhlebach M, Cies JJ, Nicolau DP, Kuti JL. Population Pharmacokinetics and Safety of Ceftolozane-Tazobactam in Adult Cystic Fibrosis Patients Admitted with Acute Pulmonary Exacerbation. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6578-6584. doi: 10.1128/AAC.01566-16. Print 2016 Nov. PMID 27550351
- [Background] Xiao AJ, Miller BW, Huntington JA, Nicolau DP. Ceftolozane/tazobactam pharmacokinetic/pharmacodynamic-derived dose justification for phase 3 studies in patients with nosocomial pneumonia. J Clin Pharmacol. 2016 Jan;56(1):56-66. doi: 10.1002/jcph.566. Epub 2015 Aug 25. PMID 26096377